CLINICAL TRIAL: NCT05712915
Title: The Extension of Rapid Response Team Operation Time and Incidence of General Ward Cardiopulmonary Resuscitation Incidence; A Retrospective Observational Study
Brief Title: Extension of Rapid Response Team Operation Time and Cardiopulmonary Resuscitation Incidence
Status: Completed | Type: Observational
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Dong Hyun Lee, professor, Dong-A University Hospital
Other Study IDs: RRT_CPR
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Cardiopulmonary Arrest
Keywords: cardiopulmonary arrest; rapid response team; operation time
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RRT operation — A retrospective observational study was conducted at a 990-bed tertiary care referral teaching hospital from April 2014 to December 2020. The RRT implemented in April 2017 as a part-time RRT operating 8 hours on weekdays. In March 2018, operation time was extended to 15 hours on weekdays and finally, extended to 24 hours a day, 7 days a week in February 2019.
  Impact of RRT operation on CPR incidence was retrospective analyzed without any prospective intervention.

SUMMARY:
Although early rapid response team was reported as a full-time operating system, similar efficacy of part-time rapid response team has been recently reported. We sought to investigate the association between the duration of rapid response team operation time and the incidence of general ward cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
Rapid response team (RRT) was introduced to reduce the preventable cardiac arrest in general wards and it has been spread worldwide. RRTs usually consist of dedicated intensivists in RRT and nurse specialists in critical care.

Although RRT implementation could useful, it is not suitable for all hospital circumstances because it is required high cost and plenty of experience in critical care settings. For this reason, to minimize the RRT operating cost, the part-time RRT operation was reported. Recently similar efficacy in part-time operation RRT was reported. However, it is difficult to compare full-time and part-time RRT and no study has been reported the efficacy according to the intensity of RRT operation time.

Authors invested the incidence of general ward cardiopulmonary resuscitation according to the RRT operation time; from the initial implementation to the full-time RRT operation after stepwise extension.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to study hospital from April 1, 2014, to December 31, 2020

Exclusion Criteria:

1. Patients who developed CPR in elsewhere not GW (ICU, emergency department, operation room, outpatient clinics, cardiac catheterization laboratory)
2. younger than 18 years
3. Patients admitted via the emergency department

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to study hospital from April 1, 2014, to December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 142088 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
General ward CPR incidence during period without RRT (rapid response team) | at the end of period of no RRT operation. (31th March, 2017)
General ward CPR incidence during period of part time RRT | at the end of part time RRT period (28th February, 2018)
General ward CPR incidence during period of extended part time RRT | at the end of extended part time RRT period (31st January, 2019)
General ward CPR incidence during period of full time RRT | at the end of full time RRT period (31th December, 2020)

CONTACTS AND LOCATIONS:
Locations (1):
- DongA university hospital, Busan, Seo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No